CLINICAL TRIAL: NCT01230450
Title: Feasibility of Comparing Two Surgical Treatment of Female Urodynamic Stress Incontinence (SITOT)
Brief Title: Feasibility of Comparing Two Surgical Treatment of Female Urodynamic Stress
Acronym: SITOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Aberdeen Royal Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI-TOT
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Female Stress Incontinence
Keywords: urodynamic urinary incontinence, sub-urethral tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-incision Mini-slings (SIMS- Ajust) (Experimental): AjustTM has polypropylene fixing anchors (one is fixed and the other adjustable) which are anchored onto the obturator membrane. The pulley like system enables adjustment of the tension once the arms have been anchored. Once in place, the anchors rest at right angles to insertion which is claimed to reduce the chances of anchor dislodgment
  Interventions: Procedure: sub-urethral tape (TVT-O)
- standared med urethral sling (SMUS) (Other): standard med urethral sling (SMUS)TVT-O, was done as originally described by Deleval et al.
  Interventions: Other: stand standard mid-urethral sling (TVT-O)

INTERVENTIONS:
Procedure: sub-urethral tape (TVT-O) — Tension free vaginal tape vs. single incision sub-urethral tension free vaginal tape
  Arms: Single-incision Mini-slings (SIMS- Ajust)
Other: stand standard mid-urethral sling (TVT-O)
  Arms: standared med urethral sling (SMUS)

SUMMARY:
Aim: The study aim to assess the feasibly a large prospective multi-centre randomised study for comparing the relatively new "Single incision sub-urethral tapes" with the standard surgical treatment of female urodynamic stress incontinence (USI).

DETAILED DESCRIPTION:
Single incision tension-free sub-urethral vaginal tapes procedures8 have been recently described in an attempt to avoid the blind passage of the trochars through the groin & the adductor muscles and consequently reducing the incidence & severity of postoperative leg pain. The obvious advantages would be shorter hospital stay, early recovery, early resumption of day to day activities & earlier return to work. A number of small prospective audits and case-series have been presented in international conferences reporting on the safety & outcomes for these procedures. However all these studies were for preliminary reports for proof of concept and therefore the studies populations were 15-70 women with short term follow-up of 2-3 month9-11.These studies have shown low perioperative complication rates: bladder injury 0-1%, vaginal erosion 1-3% & one study showing 1.3% pain at 6 weeks follow-up. The patient reported success rates were 77-93% at 2-3 month follow-up9-12.

Objectives:

1. Establish the feasibility of the "Single incision sub-urethral tapes" to be done under local anaesthesia.
2. The feasibility of randomisation to the standard surgical treatment TVT-O / TVT.
3. To compare the surgical approach in this relatively new procedure against the standard procedures as regard: Peri-operative complication rates, Postoperative pain, Time to discharge from the hospital,
4. To compare the outcomes as regard: Patient-reported cure rates, Patient satisfaction, Impact on Quality of life (QoL) and sexual function at 3 month & 1 -year follow-up. The objective cure rates will be assessed at 3 month follow-up.

Design:

A pilot prospective randomised study within participating urogynaecology units of the "Scottish Pelvic Floor Network".

ELIGIBILITY:
Inclusion Criteria:

* USI
* Mixed incontinence symptoms with predominantly bothering stress component (No DO on UDS).
* Primary Incontinence Surgery.
* BMI < 35
* Ability to understand the information leaflet and sign an informed consent form in English.
* All would have had failed or declined PFMT.

Exclusion Criteria:

* Mixed incontinence with pre-dominant OAB and/or Neurological conditions e.g. MS.
* Detrusor Overactivity on Urodynamics.
* Inability to understand English.
* Un-willing for randomisation.
* Concomitant surgery.
* Patient requiring postoperative hospital-stay for medical or social reasons

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
• Feasibility of the single incision sub-urethral tape to be done under local anaesthesia | 1 year
  * Feasibility of the single incision sub-urethral tape to be done under local anaesthesia?
  * Number of women approached and declining LA o Number of women in LA group converted to GA

SECONDARY OUTCOMES:
• Patient-reported Success rates | 1 year
  Patient-reported Success rates
  o Assessed by PGI-I "Very Much Improved/ Much Improved."

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Fattah, MRCOG, Principal Investigator — University of Aberdeen
Locations (1):
- (Grampian) Aberdeen Royal Infermary, Aberdeen, Aberdeenshire, United Kingdom

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839